CLINICAL TRIAL: NCT02661880
Title: The Role of Music in Palliative Care: A Proposal for a Rural Based Initiative in Music Based Interventions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Music in Palliative Care
Record Dates: First submitted 2016-01-19; First posted 2016-01-25 (Estimated); Last update posted 2022-11-22 (Actual); Status verified 2016-01

CONDITIONS: Improved Emotional Regulation; Improvement in Quality of Life; Symptom Relief; Preservation of Dignity; Existential Solace; Relief of Suffering; Emotional Regulation; Quality of Life; Dignity
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- listening to preferred music choices (Experimental): All patients will be invited to complete the McGill Quality of Life Questionnaire - Revised (McGill QOL-R) upon admission to the unit. The Questionnaire will not be part of the permanent medical record and the participants will remain anonymous. Afterwards participants will be asked if they would like to listen to music during their stay in the hospital. Music will be selected according to their choices from an i-Tunes playlist. Participants will be invited to listen to music at their own discretion. Prior to discharge from the hospital or after 3 days all willing participants will be again invited to complete the McGill QOL-R questionnaire.
  Interventions: Behavioral: preferred music

INTERVENTIONS:
Behavioral: preferred music — listening to preferred music choices

SUMMARY:
Current practice in larger palliative care centers offer many supportive service modalities, which are often unavailable in the rural setting. Music Therapy by experienced registered Music Therapists is an example of such a modality. The current evidence continues to grow, identifying Music Therapy's benefits to help with symptom relief as well as to improve Quality of Life in many aspects of medicine, but especially in the context of palliative care. This proposal outlines an initiative to provide music-based interventions in a rural community palliative care unit where there is limited availability to a registered Music Therapist.

DETAILED DESCRIPTION:
Study participants in the pilot phase will include patients admitted to the Aberdeen Hospital Palliative Care Unit. Patients excluded from participating would include those unwilling to participate for any reason. All patients will be invited to complete the McGill Quality of Life Questionnaire - Revised (McGill QOL-R) upon admission to the unit. The Questionnaire will not be part of the permanent medical record and the participants will remain anonymous. Afterwards participants will be asked if they would like to listen to music during their stay in the hospital. Music will be selected according to their choices from an i-Tunes playlist. Participants will be invited to listen to music at their own discretion. Prior to discharge from the hospital or after 3 days all willing patients will be again invited to complete the McGill QOL-R questionnaire. The participants will remain anonymous, but will be identified as to whether they listened or did not listen to music during their hospitalization.

ELIGIBILITY:
Inclusion Criteria:

* patients admitted to the Aberdeen Hospital Palliative Care Unit.

Exclusion Criteria:

* those patients unwilling to participate for any reason

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-03-07 (Actual); Primary Completion 2016-04-06 (Actual); Study Completion 2017-04-06 (Actual)

PRIMARY OUTCOMES:
Quality of Life-using the McGill QOL-revised questionnaire | within 3 months of data collection

CONTACTS AND LOCATIONS:
Overall Officials: Anne M Kwasnik-Krawczyk, Principal Investigator — Dalhousie University

IPD SHARING:
Plan to Share IPD: No